CLINICAL TRIAL: NCT06013631
Title: Effects of Prosthesis Training With and Without Phantom Exercises on Pain, Prosthesis Satisfaction and Ambulatory Status of Lower Limb Amputees
Brief Title: Effects of Prosthesis Training on Pain, Prosthesis Satisfaction and Ambulatory Status of Lower Limb Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-315-01-2023
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
Keywords: Phantom limb pain; Prosthesis; Prosthesis training; Prosthesis satisfaction
MeSH Terms: conditions — Wounds and Injuries; Phantom Limb

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The accessor will be unaware of treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phantom Exercises (Experimental): The phantom exercises involved visualizing and then trying to perform the movements of the phantom limb.
  1. Place the limb at the angle at which they were sensing their phantom limb.
  2. Put their healthy limb in the identical spot as they perceived their phantom limb.
  3. Move their two limbs in opposition to one another.
  4. Go back to where they started. The movements included ankle inversion and eversion, flexion and extension, and adduction and abduction with toe flexion and extension, respectively.
  5. Once the patient is at ease, movements like hip or knee flexion/extension are performed until the PLP is gone.
  6. Phantom exercises will be performed as many times as possible in a single session up to 15 times until the PLP fully subsided.
  Interventions: Other: Phantom Exercises
- Prosthesis Training (Active Comparator): Training for prostheses at the appropriate amputation level will be provided. Conventional gait training protocols include Tandem walk, within parallel bar, controlled environment, full length Mirror on one side, weight shifting, shifting onto the Prosthetic Side, Pelvic rotation, Stepping on multiple heights and positions, Tandem walk, within parallel bar, and weight shifting. Gait training will last six weeks in total.
  Interventions: Other: Prosthesis Training

INTERVENTIONS:
Other: Prosthesis Training — Training for prostheses at the appropriate amputation level will be provided. Conventional gait training protocols include Tandem walk, within parallel bar, controlled environment, full length Mirror on one side, weight shifting, shifting onto the Prosthetic Side, Pelvic 22 rotation, Stepping on multiple heights and positions, Tandem walk, within parallel bar, and weight shifting. Gait training will last six weeks in total.
  Arms: Prosthesis Training
Other: Phantom Exercises — The phantom exercises involved visualizing and then trying to perform the movements of the phantom limb.
  Arms: Phantom Exercises

SUMMARY:
The objective of the study is to assess the effects of prosthesis training with and without phantom exercises on pain, prosthesis satisfaction and ambulatory status of lower limb amputees treated with prosthesis training, phantom exercises and routine physical therapy.

DETAILED DESCRIPTION:
Amputation is a catastrophic incident in a person's life which resulted in psychological, social and physical consequences. Loss of extremity resulted in negative impact on patient's body and perception as well. Phantom limb pain (PLP) can be defined by discomfort or pain in lost part of limb experienced by lower limb amputees. Phantom limb pain is physically and mentally draining condition which affects patient's daily activities like personal care and functional independence.

Phantom limb pain is highly prevalent condition among lower limb amputees. It is associated with negative effect on mental and physical health conditions. There are studies conducted on prosthesis training for prosthesis satisfaction.

However, according to researcher knowledge effects of prosthesis training along with phantom exercises have not been measured on prosthesis satisfaction. This study will encourage future studies on this topic and will help in developing state of art treatment of phantom limb discomfort associated with lower limb subtraction. As managing phantom discomfort can result in better prosthesis satisfaction and eventually ease the ambulatory status of patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years
2. Gender: male/female
3. Unilateral lower limb amputees (trans-femoral, trans-tibial) and using prosthesis and having phantom limb pain will be included.
4. Limb deficiency and phantom limb questionnaire was used for screening of patients

Exclusion Criteria:

1. Severe systematic illness
2. Psychological issues
3. Hearing/ visual impairment
4. Malignancies
5. Infectious disease
6. Neuropathic pain except PLP and residual limb pain
7. Any disorder that restricts movement of opposed limb, limited range of motion in sound limb
8. Taking pain relief medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Prosthesis satisfaction level | It will be assessed at 6th week after the application of intervention.
  To check prosthesis satisfaction of the amputees, Trinity Amputation and Prosthesis Experience Scales (TAPES) will be used. It assesses prosthetic satisfaction on the basis of the functional, aesthetic, and weight subscales. TAPES evaluates how well people adjust to physical limitations that may have an impact on social behavior.Scores range from 5 to 25, with higher scores indicating greater levels of adjustment.
Phantom Limb Pain Intensity | Pain intensity will be assessed at baseline and any change in pain intensity will be measured at 6th week of intervention.
  To measure pain intensity, Visual Analog Scale (VAS) will be used. VAS consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be').
Ambulation Status | Ambulation status will be observed at baseline and any change will be assessed at 6th week of intervention.
  The Amputee Mobility Predictor (AMP) analyses an amputee's movement with or without a prosthesis to determine their potential for ambulation. A rapid and simple-to-use assessment instrument called the Amputee Mobility Predictor (AMP) was used to estimate the functional condition of lower-limb amputees both with and without the use of a prosthesis. AMPPRO 0-42 (47 if the assistive device is included) and AMPPRO 0-38 (43 if the assistive device is included). Higher scores indicate better mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Ahmad, PhD, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Participants data that underlies the results after de-identification
Supporting Information: Study Protocol
Time Frame: Immediately after publication
Access Criteria: Researchers who provide methodological sound proposal